CLINICAL TRIAL: NCT04134780
Title: Pilot Investigation of Ultrasound Imaging and Spectroscopy as Early Indicators of Locally- Advanced Breast Cancer Response to Neoadjuvant Treatment
Brief Title: Ultrasound Imaging and Spectroscopy as Early Indicators of Locally-Advanced Breast Cancer Response
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gregory Czarnota, Radiation Oncologist and Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 301-2014
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Ultrasound; Spectroscopy; Characterization
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This work explores the possibility of using ultrasound imaging and spectroscopy as a way of monitoring cell death, hence, tumour response to treatment. The hypothesis here is that it can be used as a way of monitoring early response to cancer treatment and predicting which patients continue on in their therapy to have a complete pathological response as a primary endpoint and tumour size decrease as a secondary endpoint. If this work is successful it could be used in the future early on in a cancer patient's treatment to predict whether or not a course of chemotherapy or radiotherapy is going to be successful. For example, in patients in which the analysis indicates a poor response the chemotherapy regimen could be changed to a more efficacious one or for those receiving radiotherapy predicted to have a poor response a radiosensitizing agent could be used to improve outcome.

DETAILED DESCRIPTION:
The primary objective in this study is to identify optimal ultrasound spectroscopy parameters that can be used as an early predictor of pathological complete or partial response in women with locally advanced breast cancer receiving treatment with chemotherapy or combined modality chemotherapy and radiotherapy. A secondary objective is to perform an inter-user variability comparison by comparing second site data analysis outcomes with central co-coordinating site data analysis. The overarching goal of this research is to transform the delivery of neoadjuvant chemotherapy using quantitative ultrasound, which is non-invasive, inexpensive and portable to assess breast cancer therapies through functional imaging, in which tumour cell death is detected. By detecting cell death early in a treatment on the order of hours to days, rather than traditional anatomical assessments that take place weeks to months after the completion of therapy, ineffective therapies could be switched to more efficacious treatments or aggressive salvage therapy which has shown to already benefit patients. This has the potential of improving survival in addition to sparing patients unnecessary side effects of treatments that may span weeks to months. The investigators will use these quantitative methods to evaluate treatments with neoadjuvant chemotherapy in women with locally advanced breast cancer. This investigation will track the spatio-temporal changes in quantitative ultrasound surrogates of treatment response during neoadjuvant chemotherapy of locally advanced breast cancer and use these parameters to adapt clinical treatment. The study specifically will expand on single- institution research underway and involve a second clinical site. Data will be independently collected and analysis carried out at that site and at the co-ordinating site for comparison evaluating technology-use feasibility and reproducibility of results.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced breast carcinoma which has not been treated with any first-line therapy and will be treated with neoadjuvant chemotherapy or neoadjuvant combined chemo-radiotherapy
2. Measurable disease by ultrasound, or MRI performed within 28 days prior to treatment
3. Eastern Co-operative Oncology Group (ECOG) Performance Status of 0 or 1
4. Life expectancy of at least 6 months
5. Patients should have the ability to understand and the willingness to sign a written informed consent document. Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia
3. Psychiatric illness/social situations that would limit compliance with study requirements
4. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women and members of all races and ethnic groups are eligible for this trial.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Measuring the rate of treatment response between the treatment groups | Up to 5 years
  Correlate changes in ultrasound backscatter parameters obtained throughout the course of treatment with pathological complete or partial response

SECONDARY OUTCOMES:
Inter-user variability comparison | Up to 5 years
  Comparing second site data analysis outcomes with central co-coordinating site data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Czarnota, PhD, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (3):
- MD Anderson, Houston, Texas, United States
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario